CLINICAL TRIAL: NCT01315327
Title: A Double-Blind, Placebo-Controlled Study of Omega-3 Fatty Acids in Children and Adolescents With Tourette's Disorder
Brief Title: Omega-3 Fatty Acids in Tourette's Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Tourette Association of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSA Omega-3
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Tourette's Disorder
Keywords: Tourette's Disorder, Obsessive-Compulsive Disorder, tics
MeSH Terms: conditions — Tourette Syndrome; Obsessive-Compulsive Disorder; Tics | interventions — Fatty Acids, Omega-3; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 Fatty Acids (Experimental): Omega-3 Fatty Acids (fish oil), flexibly titrated up to 6000 mg/day.
  Interventions: Drug: Omega-3 Fatty Acids
- Placebo (Placebo Comparator): Olive oil placebo, looks and tastes identical to active intervention.
  Interventions: Drug: Olive oil

INTERVENTIONS:
Drug: Omega-3 Fatty Acids — Omega-3 fatty acids (derived from fish oil)
  Arms: Omega-3 Fatty Acids
Drug: Olive oil — Placebo
  Arms: Placebo

SUMMARY:
This study examines the safety and efficacy of omega-3 fatty acids (fish oil) for the treatment of Tourette's Disorder.

DETAILED DESCRIPTION:
This is a 20-week, double-blind, placebo (olive oil) controlled study examining supplemental fish oil in the treatment of tic and OCD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6 through 18 inclusive
* Meet full DSM-IV diagnostic criteria for TD or chronic motor tic disorder
* Normal laboratory results, including serum chemistries, hematology, and urinalysis
* Must be able to swallow capsules.
* Must be of normal intelligence in the judgment of the investigator.
* Subjects and parents must possess an educational level, degree of understanding and command of the English language to enable them to communicate suitably with the investigator and study coordinator and to understand the nature of the study.
* Subjects and their legal representatives must be considered reliable.

Exclusion Criteria:

* Organic brain disease, for example, traumatic brain injury residua
* Meeting criteria for mental retardation as defined by the DSM-IV.
* A history of seizure disorder (other than febrile seizure).
* A Subjects with history of Sydenham's Chorea.
* Autism, schizophrenia or other psychotic disorders.
* A primary diagnosis of a major mood disorder that requires ongoing psychiatric treatment.
* A neurological disorder other than a tic disorder.
* A documented auto-immune disorder.
* A major medical illness.
* A history of ongoing or previously undisclosed child abuse (risk of removal from home would not allow for consistent caretaker ratings).
* Subjects who, in the opinion of the investigator, are unsuitable in any other way to participate in this study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2003-05; Primary Completion 2006-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | Baseline and then weekly for 20 weeks
  This assessment captures tic type and frequency as well as intensity and complexity, and impairment due to tics.

SECONDARY OUTCOMES:
Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) | Baseline and then weekly for 20 weeks
  Assesses type, frequency, and impairment of obsessions and compulsions

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Gabbay, MD, MS, Principal Investigator — NYU School of Medicine; Barbara J Coffey, MD, MS, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Child Study Center, New York, New York, United States

REFERENCES:
- [Result] Gabbay V, Babb JS, Klein RG, Panzer AM, Katz Y, Alonso CM, Petkova E, Wang J, Coffey BJ. A double-blind, placebo-controlled trial of omega-3 fatty acids in Tourette's disorder. Pediatrics. 2012 Jun;129(6):e1493-500. doi: 10.1542/peds.2011-3384. Epub 2012 May 14. PMID 22585765